CLINICAL TRIAL: NCT01705379
Title: A Multicenter, Single Arm, Post Marketing Surveillance Study to Monitor the Safety of Novartis Meningococcal ACWY Conjugate Vaccine (MenACWY-CRM) Administered According to the Prescribing Information to Healthy Subjects 2 Years of Age and Older in the Philippines
Brief Title: Safety of One Dose of Meningococcal ACWY Conjugate Vaccine in Subjects 2 Years of Age and Older
Status: Withdrawn | Type: Observational
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: V59_45OB
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Meningococcal Disease
Keywords: Neisseria meningitidis, conjugate vaccine, phase IV clinical trial
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MenACWY-CRM: 2 years of age and older
  Interventions: Biological: Novartis Meningococcal ACWY Conjugate Vaccine

INTERVENTIONS:
Biological: Novartis Meningococcal ACWY Conjugate Vaccine — Immunization

SUMMARY:
A multicenter, single arm, postmarketing surveillance study. This study is a postlicensure requirement of the Philippine Food and Drug Administration (FDA) to provide continued safety evaluation of MenACWY-CRM in Philippine individuals 2 years of age and older, receiving MenACWY-CRM vaccination according to routine clinical practice and prescribing information.

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible for enrolment in this study are those:

1. who are of any gender, from the age of 2 and older, and to whom/whose parents or legally acceptable representatives the nature of the study has been described and the subject/subject's parent/legally acceptable representative has provided written informed consent.
2. who the investigator believes that the subject and/or his or her parent/legal representative can and will comply with the requirements of the protocol.
3. who are in good health as determined by clinical judgment of the investigator.

Exclusion Criteria:

Individuals not eligible to be enrolled in the study are those:

1. who are unwilling or unable to give written informed consent or assent to participate in the study.
2. who are perceived to be unreliable or unavailable for the duration of the study period.
3. who have previously been immunized with a meningococcal vaccine or vaccine containing meningococcal antigen(s) (licensed or investigational).
4. who have received any investigational or non-registered product (drug or vaccine) within 30 days prior to enrolment or who expect to receive an investigational drug or vaccine prior to the completion of the study.
5. who have received or who are planning to receive any vaccines (other than routine childhood vaccines) within 30 days before and after administration of study vaccine.

   (Exception: Influenza vaccine may be administered up to 15 days prior to study vaccination and at least 15 days after study vaccination)
6. who have behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
7. who are pregnant or breast feeding (female subjects of appropriate age) or who plan to become pregnant during the course of the study.
8. who have any serious acute, chronic or progressive disease (e.g., any history of neoplasm, cancer, diabetes, cardiac disease, autoimmune disease, HIV infection or AIDS, or blood dyscrasias, with signs of cardiac or renal failure or severe malnutrition), who have epilepsy or any progressive neurological disease or history of Guillain-Barre syndrome.
9. who have a history of any anaphylaxis, serious vaccine reactions, or allergy to any vaccine components.
10. who are known to have a bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
11. who are included in study personnel or close family members of personnel conducting this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy male and female subjects 2 years of age and older
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
All adverse events | Day 29
All serious adverse events | Day 29